CLINICAL TRIAL: NCT05066412
Title: A Phase I Clinical Trial Assessing Prophylactic Donor CD45RA-depleted Lymphocyte Infusions Into Patients Transplanted with Stem Cell Grafts from Haploidentical Donors After Reduced Intensity Conditioning
Brief Title: Prophylactic CD45RA-depleted DLI After Haploidentical Transplantation/RIC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Anne-Claire Mamez, Principal Investigator, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cd45RA depleted DLI
Record Dates: First submitted 2021-07-09; First posted 2021-10-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Hematologic Malignancy; Haplo-identical Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Prophylactic CD45RA-depleted DLI
  Interventions: Other: CD45RAneg cells, prepared from mononuclear cell leukapheresis by CliniMACS® technology

INTERVENTIONS:
Other: CD45RAneg cells, prepared from mononuclear cell leukapheresis by CliniMACS® technology — CD45RAneg cells, prepared from mononuclear cell leukapheresis by CliniMACS® technology

SUMMARY:
To assess safety of prophylactic escaladed dose of T naïve depleted (CD45RA depleted donor lymphocyte infusion, in patients with malignant hemopathie who received an allogeneic stem cell transplant from an haplo-identical donor, after a reduced intensity conditionning regiment.

DETAILED DESCRIPTION:
Primary Objective is to determine whether the administration of prophylactic CD45RAneg (CD45RAneg) memory/effector T lymphocytes is feasible and safe in the early post-transplant period for patients with haploidentical transplant and RIC conditioning.

Donor lymphocytes are isolated from the original donor by non-mobilized mononuclear cell leukapheresis. Repetitive intravenous infusions (up to 3) of escalating doses of CD45RAneg cells, prepared from the leukapheresis by CliniMACS® technology (CD45RA-depletion), storage in vapor nitrogen.

Escalating doses of CD45RAneg cells, for patients with haploidentical graft, intervals of 6-8 weeks, if GvHD is absent starting ≥ 4 weeks from the day of transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a stem cell graft from a haploidentical donor after RIC for hematologic malignancies
* Written informed consent of patient and donor obtained

Exclusion Criteria:

* Participant taking Prednisone (or equivalent steroid)
* Participant taking Prednisone (or equivalent steroid)
* Participant taking Mycophenolate Mofetil
* Participant taking Cyclosporine/tacrolimus at therapeutic blood levels
* Progressive hematologic malignancy before transplant
* Second allogeneic transplant
* Acute GvHD ≥ grade 2
* Chronic moderate or severe GvHD (NIH consensus criteria)
* Hematologic or molecular relapse of the primary malignancy requiring chemotherapy or unmanipulated DLI (receiving prophylactic antileukemic agent, eg TKI, is not an exclusion criteria)
* Donor aberrant CD45RA expression due to a polymorphism in CD45 gene
* Participation in another interventional clinical trial within 30 days prior to inclusion
* Pregnant or nursing women. Sexually active women with childbearing potential as well as sexually active male patients who are unwilling to use an effective method of contraception during participation in the study from time of inclusion until 2 months after last dose of CD45RAneg DLI infusion
* Inability to follow the procedures of the study, including, but not limited to, language problems, psychological disorders, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
acute transfusion reaction (CTCAE ≥ 2) | 24 hours after each CD45RA neg DLI infusion
  acute transfusion reaction after each DLI infusion (CTCAE ≥ 2)
acute GvHD grade II-IV | within 8 weeks after each CD45RAneg DLI infusion
  acute GvHD grade II-IV measured with MAGIC score

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No